CLINICAL TRIAL: NCT03746379
Title: Investigation of the Relationship Between Sensory Processing and Kinesychophobia in
Brief Title: Investigation of the Relationship Between Sensory Processing and Kinesychophobia in Fibromyalgia Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Principal Investigator, Trakya University
Other Study IDs: 2018/359
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Fybromyalgia
Keywords: kinezyhophobia; sensory processing; fybromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fibromyalgia; is a chronic and rheumatic condition characterized by diffuse pain. In patients with fibromyalgia syndrome, there is an increase in psychiatric symptoms, especially depression, anxiety, and somatoform disorders. Kinesophobia is defined as anxiety against pain and pain caused by painful injury and re-injury. The aim of this study was to investigate the relationship between kinesophobia and sensory processing in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia; is a chronic and rheumatic condition characterized by diffuse pain. In patients with fibromyalgia syndrome, there is an increase in psychiatric symptoms, especially depression, anxiety, and somatoform disorders. Kinesophobia is defined as anxiety against pain and pain caused by painful injury and re-injury. The aim of this study was to investigate the relationship between kinesophobia and sensory processing in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Diagnosed by fibromyalgia
* No other known physical, neurological and psychological illness
* Literate
* Volunteers to participate in the study

Exclusion Criteria:

* Not compliant with inclusion criteria

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2018-12-16 (Estimated); Primary Completion 2019-01-17 (Estimated); Study Completion 2019-02-18 (Estimated)

PRIMARY OUTCOMES:
Sensory processing assessed with the Sensory Adolescent / Adult Sensory Profile Questionnaire | at the end of the third month
  Sensory processing disorder refers to the difficulty of processing the information coming from the sensory organs, and the inefficiency of the normal sensory processing process.For the evaluation of sensory processing; Sensory Adolescent / Adult Sensory Profile questionnaire will be used.
Knesychophobia assessed with the Tampa Kineshiophobia Scale | at the end of the third month
  Kinezyophobia is defined as anxiety against pain and pain caused by painful injury and re-injury. For the evaluation of kinesiophobia; Tampa Kineshiophobia Scale will be used.

IPD SHARING:
Plan to Share IPD: Undecided